CLINICAL TRIAL: NCT04942366
Title: Effects of High-Intensity Interval Training and Strength Training On Levels of Testosterone and Physical Activity Among Women With Polycystic Ovary Syndrome.
Brief Title: High-Intensity Interval Training On Women With Polycystic Ovary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Mubarra Rao, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mubarra Rao
Record Dates: First submitted 2021-06-19; First posted 2021-06-28 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: High intensity interval training; Exercise; Polycystic Ovary Syndrome; Physical Therapy; Strength training; Testosterone; Physical activity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Intervention Model Description: Two groups in which participants are randomly allocated while both groups will perform warm up and cool down session, Group A will perform High intensity interval training and Group B will perform strength training exercises.
Who Masked: Participant, Care Provider
Masking Description: While the exercise protocol will be explained to the participant and care giver however the they will be blinded regarding which is intervention group or control group and which exercise is the main interventional exercise will not be disclosed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Group (Experimental): High intensity interval training will be performed thrice a week using a treadmill.
  Interventions: Other: High intensity interval training
- ST Group (Active Comparator): Strength training will be performed thrice a week, each session will consist of eight dynamic drills (with resistance of 60 - 70 % of 1 repetition maximum).
  Interventions: Other: Strength training

INTERVENTIONS:
Other: High intensity interval training — HIIT using treadmill four sets of 4 minute interval session (at 90%-95% of the individual HR max calculated by using the karvonen method) and each set will be followed by three minute of moderate intensity exercise (at 70% of individual HR max).
  Other Names: HIIT
  Arms: HIIT Group
Other: Strength training — Strength training will be performed thrice a week, each session will consist of eight dynamic drills.
  Arms: ST Group

SUMMARY:
This RCT is aimed towards determining the effectiveness of exercises based intervention strategy involving high intensity interval training exercises in improving serum testosterone level, body fat composition and physical activity in hopes to provide a definitive exercise regime for the ever common symptoms of pcos. It will be based on the theory that exercise helps in decreasing testosterone level that in turn decrease high androgen levels in the body, exercise further decreases body fat composition (obesity is a common cause or manifestation of pcos).

DETAILED DESCRIPTION:
High intensity interval training will be performed over the course of 12 weeks and will be compared with the group performing strength training. Baseline assessments will be done before the start of the first session and post-test assessment will be done after the last session of the study.

Envelope method is used for the purpose of randomization. 50 envelopes having a title of group A and group B will be made and divided into two (25 in each group). Mutually exclusive technique will be used and the envelope once picked will not be replaced within the groups.

Sample size is calculated by using a previous study conducted in 2015 titled as, 'Effects of High Intensity Interval Training and Strength Training on Metabolic, Cardiovascular and Hormonal Outcomes in Women with Poly cystic Ovary Syndrome: A Pilot Study' by taking a confidence interval CI of 95%, power of test 80%, standard deviation of 6.3 and mean difference of 5.2, a sample size of 50 is calculated.

For the analysis of the data MedCalc software version 19.0.5. will be used. Descriptive statistics will be performed for the purpose of demographic information and this data will be presented in terms of frequency and percentage. Skewness and Kurtosis will be used in order to determine the normality of data. If the data is normally distributed, then for within the group analysis dependent T test will be performed. However, in case the data is not normally distributed Wilcoxon Sign Rank test will be performed. Independent T test will be performed for the comparison between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI:

  1. Overweight: 23-24.9 kg/m2.
  2. Obese: greater than or equal to 25 kg/m2 .
* Diagnosed and referred PCO patients to the rehabilitation unit would be selected for the study.
* Aged 18-40.
* High serum testosterone level: normal range 6-86 ng/dl.

Exclusion Criteria:

* On-going pregnancy.
* Any cardiovascular complication.
* Any other endocrine disorder
* Any musculoskeletal condition that hinders in performing the exercise training protocol.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mubarra Rao, Principal Investigator — Ziauddin University; Amna Amir Khan, Study Director — Ziauddin University
Locations (1):
- Shamim clinic, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Serum testosterone was more than normal. Pre-diagnosed PCOS. Overweight or/and obese. Physical activity level (IPAQ).
Period: Overall Study
Arm/Group | HIIT Group | ST Group
Started | 25 (5 withdrew from the study before the first session.) | 25 (5 withdrew from the study before the first session.)
Completed | 20 (5 withdrew from the study before the first session.) | 20 (5 withdrew from the study before the first session.)
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIIT Group | ST Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (4.92) | 30.5 (4.80) | 29.3 (4.86)
Sex/Gender, Customized [Number; unit: participants] — Population: 10 participants withdrew from the study, five from each group and this is the reason why at the end of the study 40 participants were analyzed.
  participants
    Females | 20 | 20 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Serum Testosterone [Mean (Standard Deviation); unit: nmol/L] — Population: Five participants withdrew from the study, this is the reason why at the end of the study 20 participants were analyzed.
  nmol/L | 2.54 (0.07) | 2.54 (0.09) | 2.54 (0.08)
Body fat percentage [Mean (Standard Deviation); unit: percentage] — Population: Five participants withdrew from the study, this is the reason why at the end of the study 20 participants were analysed.
  percentage | 31.6 (1.79) | 34.1 (2.70) | 32.9 (2.60)

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone
Description: Levels of serum testosterone
Time Frame: 0 weeks to 12-weeks
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | HIIT Group | ST Group
Number analyzed (Participants) | 20 | 20
nmol/L
  0-week | 2.54 (0.07) | 2.54 (0.09)
  12-weeks | 2.39 (0.14) | 2.47 (0.09)

2. Primary Outcome: Body Fat Percentage
Description: Using skinfold method (body caliper)
Time Frame: 0-week to 12-weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | HIIT Group | ST Group
Number analyzed (Participants) | 20 | 20
Percentage
  0-week | 31.59 (1.79) | 34.12 (2.69)
  12-weeks | 29.62 (1.76) | 32.48 (2.87)

3. Primary Outcome: Physical Activity
Description: International physical activity questionnaire
Time Frame: 0-week to 12-weeks
Measure: Mean (Standard Deviation); unit: MET-mins/week
Arm/Group | HIIT Group | ST Group
Number analyzed (Participants) | 20 | 20
MET-mins/week
  0-week | 3491.15 (211.99) | 3439.60 (243.76)
  12-weeks | 3928.10 (220.04) | 3716.60 (234.45)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | HIIT Group | ST Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04942366/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04942366/SAP_001.pdf